CLINICAL TRIAL: NCT06235229
Title: A Phase I/II Clinical Study of Chimeric Antigen Receptor T-cell Therapy Targeting CD19 and BCMA (GC012F) in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study of GC012F in Patients With Relapsed/Refractory Multiple Myeloma
Acronym: DURGA-3
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8315C00001; GBF-311 (Other: Gracell)
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Relapsed/Refractory Multiple Myeloma; Chimeric Antigen Receptor - T(CAR-T); Dual Targets; B-cell Maturation Antigen(BCMA); Cluster of Differentiation - 19(CD19)
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC012F (Experimental): GC012F will be administered by infusion
  Interventions: Biological: GC012F

INTERVENTIONS:
Biological: GC012F — GC012F is a BCMA/CD19 dual CAR product

SUMMARY:
This study is a single-arm, open-lable, phase I/II study to evaluate the efficacy and safety of GC012F in subjects with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
A leukapheresis procedure will be performed on eligible subjects to manufacture GC012F.Subjects will receive an infusion of GC012F at specified doses after three consecutive days of lymphodepletion consisting of fludarabine and cyclophosphamide. Bridging therapy is allowed between leukapheresis and lymphodepletion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of active multiple myeloma as defined by the updated IMWG (International Myeloma Working Group) criteria, and meet one or more of the following criteria:

   1. Serum M protein ≥ 1 g/dL；
   2. Urine M protein ≥ 200 mg/24hrs;
   3. Serum free light chain (sFLC) ≥ 10 mg/dL with abnormal sFLC κ/λ ratio.
2. Have received at least 3 prior lines of therapy for multiple myeloma. Note: According to IMWG guidelines, a single line of therapy includes a full course of monotherapy, combination therapy with multiple drugs, or sequential treatment with multiple regimens (e.g., the use of a 3-6 cycle regimen of bortezomib combined with dexamethasone, followed by stem cell transplantation, consolidation therapy, and lenalidomide maintenance therapy, is considered a single line of therapy). Unless the best response was documented as progressive disease (PD) or the subject was intolerant to the therapy.
3. Prior therapy should include proteasome inhibitors (PIs), immunomodulatory drugs (IMiDs), and anti-CD38 antibodies.
4. Evaluated by investigator based on IMWG standards, subjects have a confirmed (through testing at a central or local laboratory) PD during or within 12 months following the most recent anti-myeloma treatment.
5. Voluntarily signed a written informed consent form (ICF).
6. The signing of ICF complies with the requirements of GCP and relevant national laws and regulations.
7. Males or females, aged 18-75 years old (including the thresholds).
8. Subjects should be willing and able to comply with the study visit schedule and other protocol requirements.
9. ECOG (Eastern Cooperative Oncology Group) performance score 0-1.
10. Estimated life expectancy ≥ 3 months.
11. Adequate functional reserve of organs:

    1. Neutrophil count ≥ 0.75×10^9/L (growth factor support is allowed, but no supportive treatment is allowed within 7 days prior to screening); Hemoglobin ≥ 8.0 g/dL (no red blood cell transfusion within 7 days prior to screening, recombinant human erythropoietin is allowed); Platelet count ≥ 50×10^9/L (no platelet transfusion within 7 days prior to screening); Lymphocyte count ≥ 0.3×10^9/L;
    2. ALT/AST ≤ 3× ULN (upper limit of normal); Total bilirubin ≤ 2× ULN (in subjects with Gilbert syndrome, direct bilirubin ≤ 1.5× ULN is required);
    3. Creatinine clearance ≥ 40 mL/min, calculated by Cockcroft-Gault;
    4. Left ventricular ejection fraction (LVEF) ≥ 45% with no evidence of pericardial effusion as diagnosed by echocardiography; No clinically significant electrocardiogram abnormality observed;
    5. Baseline oxygen saturation ≥ 95% on room air; No clinically significant pleural effusion observed.
12. Female subjects with fertility must:

    1. Have a negative serum beta-human chorionic gonadotropin (β-hCG) pregnancy test confirmed by investigators during screening and before undergoing lymphodepletion with cyclophosphamide and fludarabine.
    2. Agree and be able to use effective contraception continuously from screening to at least 1 year after GC012F infusion. Contraception must include one highly effective and one additional effective (barrier) method, initiated from screening until at least 1 year after GC012F infusion or until two consecutive flow cytometry tests show the absence of CAR-T cells (whichever occurs later).
    3. Agree to avoid breastfeeding during the study period until at least 1 year after GC012F infusion or until two consecutive flow cytometry tests show the absence of CAR-T cells (whichever occurs later).
13. Male subjects must agree to use condoms during sexual contact with pregnant females or females with fertility for at least 2 year after GC012F infusion, even if a successful vasectomy has been performed.
14. Sufficient venous access for leukapheresis collection, and no other contraindications to leukapheresis.

Exclusion Criteria:

1. Prior treatment with CAR-T products for any target.
2. Have any of the following concomitant treatment history:

   1. Received a total of ≥ 70 mg of prednisone or an equivalent dose of other corticosteroids within 7 days prior to leukapheresis;
   2. Investigators believe that patients has comorbidities requiring the systemic use of corticosteroids (a total of ≥ 70 mg of prednisone or an equivalent dose of other corticosteroids) or other immunosuppressive drugs within 12 weeks after the start of the study treatment;
   3. Received a live-attenuated vaccine within 4 weeks prior to leukapheresis or lymphodepletion;
   4. Received any anticancer therapy, including but not limited to radiation therapy, cytotoxic therapy, PIs, IMiDs, targeted therapy, epigenetic therapy, or experimental drug treatment, within 14 days prior to leukapheresis (if radiation field covers ≤ 5% of bone marrow, subjects can be enrolled regardless of the end date of radiation therapy);
   5. Received monoclonal antibody for treating multiple myeloma within 21 days prior to leukapheresis.
3. Patients' corticosteroid maintenance doses are greater than physiological replacement doses (i.e., prednisone ≥ 7.5 mg/day or hydrocortisone ≥ 12 mg/m^2/day).
4. Patients with any of the following heart diseases:

   1. Congestive heart failure (NYHA classification ≥ III);
   2. Experienced myocardial infarction or underwent coronary artery bypass grafting (CABG) within 6 months prior to screening;
   3. Clinically significant ventricular arrhythmias or a history of unexplained syncope not due to vasovagal reaction or dehydration; or a QTc interval > 480 ms during screening;
   4. History of severe non-ischemic cardiomyopathy.
5. Patients requiring assisted oxygenation or mechanical ventilation or with oxygen saturation <95% on room air (patients with oxygen saturation <95%, but with lung function test results showing carbon monoxide diffusing capacity and forced expiratory volume in 1 second > 45% of predicted value, may be enrolled).
6. Patients with hypertension that is uncontrolled by drug therapy.
7. Patients with clinically significant bleeding symptoms or definite bleeding tendencies (e.g., gastrointestinal bleeding, bleeding gastric ulcers, etc.), hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophilia, coagulation disorders, hypersplenism, etc.) within 90 days prior to screening; have experienced arteriovenous thrombotic events (e.g., cerebrovascular diseases (including cerebral hemorrhage, cerebral infarction, etc.), deep vein thrombosis, and/or pulmonary embolism) within 180 days prior to screening.
8. Accompanied by other uncontrolled malignancies. The following are excluded: early-stage tumors that have received radical treatment (carcinoma in situ or grade 1 tumors, or non-ulcerated primary melanoma with a depth < 1 mm and no involvement of lymph nodes), basal cell skin cancer, squamous cell skin cancer, cervical carcinoma in situ, or breast carcinoma in situ that has received potential radical treatment.
9. Have received any of the following treatments:

   1. Received an allogeneic hematopoietic stem cell transplantation (allo-HSCT) within 6 months prior to leukapheresis. Patients undergoing allo-HSCT who have discontinued all immunosuppressive drugs for 6 weeks prior to leukapheresis and have no manifestations of graft-versus-host disease (GVHD) may be enrolled.
   2. Received an autologous hematopoietic stem cell transplantation (auto-HSCT) within ≤ 12 weeks prior to leukapheresis.
10. Severe underlying medical conditions, such as:

    1. Evidence of active viral or bacterial infection (requiring systemic antimicrobial therapy) or uncontrolled systemic fungal infection;
    2. Active autoimmune diseases or a history of autoimmune disease within the past 3 years;
    3. Significant clinical evidence of dementia or altered mental status;
    4. History of any central nervous system (CNS) or neurodegenerative diseases, (e.g., epilepsy, seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, psychiatric disorders).
11. Patients have CNS metastases or CNS involvement (including cranial neuropathies or mass lesions and leptomeningeal disease).
12. Positive results in any of the following tests:

    1. HIV antibody positive;
    2. HBsAg positive; or HBcAb positive, with HBV DNA titer higher than the lower limit of detection;
    3. HCV antibody positive, with HCV RNA titer higher than the lower limit detection; or known history of Hepatitis C, but did not complete antiviral treatment for ≥24 weeks;
    4. Syphilis antibody positive.
13. Accompanied by plasma cell leukemia (peripheral blood plasma cells > 2.0×10^9/L), Waldenstrom macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy of undetermined significance, skin changes), or primary amyloidosis.
14. Patients have a history of severe hypersensitivity or allergy.
15. Contraindication or hypersensitivity to fludarabine, cyclophosphamide, and any component of experimental product.
16. Surgery plan within 2 weeks prior to leukapheresis or during the study (except for local anesthesia surgery, but not performed within 2 weeks after CAR-T infusion).
17. Pregnant or lactating, or planning to have a pregnancy during or within 2 year after treatment.
18. Acute toxicities (except for hematological toxicities and alopecia) caused by previous treatments have not recovered to ≤ grade 1.
19. Participated in other clinical trials within 4 weeks prior to ICF signing, or ICF signing date is within 5 half-lives of the drug from the last medication in the last drug clinical trial (whichever is longer).
20. Any situation in which investigators believe that participation in this study is not in the subject's best interests, or any situation that may hinder patients' participation in the entire trial or confuse the assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Dose-limiting toxicities | 28 days post GC012F infusion
  The incidence of DLT within 28 days post infusion
Phase 2: Overall response rate | Minimum of 2 year post GC012F infusion
  Overall response rate according to IMWG 2016

SECONDARY OUTCOMES:
Adverse events | Minimum of 2 year post GC012F infusion
  The incidence and severity of adverse events
Pharmacokinetics: Cmax | Minimum of 2 year post GC012F infusion
  The maximum trangsgene level at Tmax
Pharmacokinetics: Tmax | Minimum of 2 year post GC012F infusion
  Time to peak transgene level
Overall survival (OS) | Minimum of 2 year post GC012F infusion
  Time from GC012F infusion to the date of death due to any cause
Duration of response (DOR) | Minimum of 2 year post GC012F infusion
  Time from initial response to the date of disease progression
Progression-free survival (PFS) | Minimum of 2 year post GC012F infusion
  Time from GC012F infusion to the date of disease progression
Minimal residual disease (MRD) | Minimum of 2 year post GC012F infusion
  Proportion of subjects who achieved MRD negative

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Research Site, Beijing
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/